CLINICAL TRIAL: NCT00271063
Title: Phase I/II Study of Liposomal Annamycin in Patients With Refractory or Relapsed Acute Lymphocytic Leukemia
Brief Title: Study of Liposomal Annamycin in Patients With Refractory or Relapsed Acute Lymphocytic Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Callisto Pharmaceuticals (Industry)
Responsible Party: Gary Jacob, Callisto Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-103
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Acute Lymphocytic Leukemia
Keywords: Refractory or Relapsed Acute Lymphocytic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Liposomal Annamycin — 3-day IV infusion

SUMMARY:
This is a Phase I/II multi-center, open label, dose escalation study to identify the maximum tolerated dose (MTD) of liposomal annamycin and to evaluate the safety of liposomal annamycin in patients with refractory or relapsed acute lymphocytic leukemia.

DETAILED DESCRIPTION:
This is a Phase I/II, multi-center, open-label, dose escalation, MTD study of liposomal annamycin in refractory or relapsed ALL patients. Enrollment will occur in cohorts of approximately 3 patients with 10 additional patients enrolled at the MTD. The liposomal annamycin doses will be escalated in sequential cohorts. Four dose levels of liposomal annamycin are planned: 190, 230, 280, and 310 mg/m2/day.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of refractory or relapsed ALL (acute lymphocytic leukemia)
* Age greater than or equal to 15 years
* No chemotherapy, radiation, or major surgery within 2 weeks prior to first dose of study drug and recovered from toxic side effects of that therapy, unless treatment is indicated due to progressive disease.
* No investigational therapy within 4 weeks of first dose of study drug
* ECOG performance status (PS) 0 to 2.
* Adequate liver function
* Adequate renal function
* Signed informed consent

Exclusion Criteria:

* Concommitant therapy that includes other chemotherapy that is or may be active against ALL (except central nervous system [CNS] therapy)
* Any condition which in the opinion of the investigator, places the subject at unacceptable risk if he/she were to participate in the study.
* Cardiac ejection fraction less than 40%
* Clinically relevant serious co-morbid medical conditions.
* Pregnant, lactating or not using adequate contraception.
* Known allergy to doxorubicin or anthracyclines.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2005-10; Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of L-Annamycin | 8 months
MTD | 8 months

SECONDARY OUTCOMES:
To study multi drug-resistant (MDR)-1 encoded P-170 glycoprotein expression and MDR-1 multidrug-resistant-associated protein (MRP), lung-resistance associated protein LRP), and breast cancer resistance protein (BCRP) mRNA levels | 8 months
To measure the pharmacokinetics of annamycin and its metabolite, annamycinol. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary Jacob, PhD, Study Director — Callisto Pharmaceuticals
Locations (3):
- United States (3):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Montefiore Medical Center, The Bronx, New York
  - MD Anderson Cancer Center, Houston, Texas